CLINICAL TRIAL: NCT03720223
Title: Liposomal Bupivacaine To Control Post-Operative Pain Following Buccal Mucosal Graft Harvesting
Brief Title: Liposomal Bupivacaine To Control Post-Operative Pain Following BMG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urology of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-09-FB-0185
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Urethral Stricture
Keywords: Buccal mucosal graft
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient blinded for the intraoperative intervention given (With Liposomal Bupivacaine injection to the buccal mucosal graft harvest site or not)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine (Experimental): 20ml Liposomal Bupivacaine 1.3% (13.3mg/mL), injected to the buccal mucosal graft harvest site.
  Interventions: Drug: Liposomal Bupivacaine
- Control (No Intervention): No local anesthetics injected to the buccal mucosal graft harvest site

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 20ml of Liposomal Bupivacaine 1.3% (13.3mg/mL)
  Other Names: Exparel
  Arms: Liposomal Bupivacaine

SUMMARY:
This is a single blinded-randomized controlled trial that recruit male patients for substitution urethroplasty using buccal mucosal graft. The study investigators aim to assess the efficacy and safety of liposomal bupivacaine injection to the buccal graft harvest site on post-operative main score, morphine equivalence requirement and oral morbidities.

DETAILED DESCRIPTION:
Pain following urethroplasty with buccal mucosal graft (BMG) harvesting is primarily related to the oral graft harvest site. This pain results in significant increases in narcotic use, patient morbidity, and limits nutritional intake following surgery. During BMG harvesting, lidocaine with epinephrine is routinely injected for hydrodissection and to assist with hemostasis. The analgesic benefits from this local anesthetic, however, have abated prior to completion of the urethral reconstruction and contribute little to post-operative pain control.

In an effort to alleviate pain following BMG harvesting, several centers have evaluated technical aspects of the procedure to reduce post-operative pain. These have primarily focused on location of the graft harvest and wound closure. A novel liposomal formulation of bupivacaine has recently been introduced as a 96-hour delayed release formulation. It has been safely used in multiple surgical wounds and results in significantly reduced post-operative pain and narcotic usage. Given that patient reported pain from the BMG harvest site is worst in the first 1-2 days following surgery, infiltration of this medication has the potential to dramatically reduce post-operative pain in these patients.

Objectives:

Our objective is to evaluate post-operative pain and narcotic usage following BMG harvesting with liposomal bupivacaine infiltration. Our hypothesis is that infiltrating the buccal graft harvest surgical site with liposomal bupivacaine will decrease both post-operative pain and narcotic usage and increase patient satisfaction.

Study Design:

The study will be a prospective, randomized, single blind controlled trial. Patients will be recruited from the offices of Urology of Virginia, Devine-Jordan Center for reconstructive surgery and pelvic health. Eligible patients will include all males 18 years of age or older identified as requiring a urethroplasty with BMG harvesting. On the initial visit, eligible patients will complete a research consent.

Patients will be randomized to receive either standard of care BMG harvesting or standard of care plus buccal infusion of liposomal bupivacaine. Randomization will be determined with a random number generator in the Urology of Virginia research office prior to surgery. Patient randomization will be revealed to the operative surgeon on the day of surgery following induction of general anesthesia. The remainder of the procedure will be performed as per routine.

Post-operatively, a member of the research team who was not a member of the operative team will monitor the patient's pain and narcotic usage. Pain will be assessed using a validated 10-point pain scale as well as a non-validated BMG harvest site morbidity questionnaire, an evaluation technique that has been used previously. Inpatient narcotic usage will be calculated post-op through cumulative morphine equivalents on a 24-hour basis on the day of surgery as well as post-op days one, two and three. All patients are routinely discharged home on post-op day two or three. The pain and morbidity questionnaire will be administered in the pre-operative holding area, then daily for the first seven days followed by monthly through 6 months of follow up. Studies have shown a return to baseline pain within six months following BMG harvesting and assessments beyond that time are unnecessary. Responses to questionnaires will be obtained either by a member of the Urology of Virginia research staff through either a phone call or email message to the patients at each time point. Preferred method of contact, including a preferred phone number and email address will be obtained during the initial visit when study consent is obtained.

The primary endpoint will be reduction in post-op pain on the 10-point numerical rating scale, post-operative narcotic requirements and oral morbidities. Secondary endpoints will be return of eating a regular diet, perioral numbness, salivary changes and the ability to open the mouth completely.

Power analysis shows that 40 patients would be required to attain 80% power to detect a > 1 point change in the numeric pain scale at a 2-sided level of 5%. Accounting for 10-20% dropout rate, the study investigators plan to recruit 50 patients for randomization.

The Urology of Virginia research department will maintain all study data. Patients will be identified by medical record number for the purpose of data collection. However, in the database, patient information will be associated only with a non-identifying subject identification number that will be assigned at study entry. A file linking patient medical record numbers with subject identification numbers will be maintained separately from the database. All files will be kept on an encrypted, password-protected external data drive for additional security. All files will be destroyed no later than three years following the end of the study.

Safety monitoring for this study will be done at each subject encounter and maintained within the Urology of Virginia research office. Adverse effects will be queried during each interaction with the patient and is also included in the questionnaire to be filled out throughout the study period.

Rudimentary statistical analysis will be carried out using excel spreadsheets, which will include mean/median values, percentages and data trends. Additionally, multivariate regressions models will be created using the Statistical Package for the Social Sciences (SPSS) software.

Risk to Subjects:

Liposomal bupivacaine has been used for several years in a variety of surgical settings without significant adverse events compared to traditional bupivacaine. However, its specific use in buccal infiltration for BMG harvesting has not previously been reported.

Liposomal bupivacaine has been studies in several clinical trials. The reported adverse reactions related to its use include, but are not limited to:

* Most common

  o Nausea, constipation, and vomiting.
* Common

  o Fever, dizziness, peripheral swelling, anemia, hypotension, pruritus, tachycardia, headache, insomnia, muscle spasms, back pain, somnolence, and procedural pain.
* Less common/rare

  o Chills, erythema, bradycardia, anxiety, urinary retention, pain, edema, tremor, dizziness postural, paresthesia, syncope, incision site edema, procedural hypertension, procedural hypotension, procedural nausea, muscular weakness, neck pain, pruritus generalized, rash pruritic, hyperhidrosis, cold sweat, urticaria, bradycardia, palpitations, sinus bradycardia, supraventricular extrasystoles, ventricular extrasystoles, ventricular tachycardia, hypertension, pallor, anxiety, confusional state, depression, agitation, restlessness, hypoxia, laryngospasm, apnea, respiratory depression, respiratory failure, body temperature increased, blood pressure increased, blood pressure decreased, oxygen saturation decreased, urinary retention, urinary incontinence, vision blurred, tinnitus, drug hypersensitivity, and hypersensitivity.
* Specific neurological and cardiac adverse reactions o Dizziness (6.2%), headache (3.8%), somnolence (2.1%), hypoesthesia (1.5%), and lethargy (1.3%), tachycardia (3.9%) and bradycardia (1.6%).

This study does involve data collection from medical records and depends upon patient identifiers for data collection. HIPAA compliance in clinical data handling will ensure protection of patient's right to privacy. Information in the database will be non-identifiable. All collected data will be stored on an encrypted, password-protected external data drive. No personal health information data will be released. Only investigators listed within this Institutional review board proposal will have access to the data collected. Despite these safeguards, there is always risk for incidental release of patient personal health information. As outlined above, every effort will be made to limit these risks.

Disposition of Results:

The results of this study will be communicated in presentations at society meetings (such as the American Urologic Association national meeting). Final disposition of this study will be submitted for publication in a peer-reviewed scientific journal. All information is unidentified.

ELIGIBILITY:
Inclusion Criteria:

* male adults with urethral stricture assessed to be requiring a urethroplasty with BMG harvesting

Exclusion Criteria:

* female adult patient with urethral strictures
* prior diagnosis of chronic pain or systemic disease that would interfere with outcome assessment or metabolism of the local anesthetics or narcotics.
* allergy to liposomal content or bupivacaine or any cross reaction to local anesthetics
* neurological disease with impaired communication or neurological deficit to pain
* with poor oral health with lesions
* urethroplasties with no requirement for BMG graft
* on daily narcotic requirement pre-operatively
* on daily analgesia medication required for other condition
* consented for other clinical trials which may interfere the outcome assessment
* unwilling for post-operative interview or survey involvement

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain score | Post-op day 1
  Continuous variables to be assessed as: Post-operative oral pain score measured using 10 point visual analogue score for pain assessment (minimum 0 or no pain to maximum 10 most painful)
Morphine equivalent requirements | Post-procedure day 1
  Continuous variable to be assessed as : Narcotics requested by the patient and administered post-procedural day 1 and day 2 (Total and separately assessed). All narcotics will be converted to IV morphine equianalgesic equivalent conversion factors according to American Pain Society
Morphine equivalent requirements | post-procedure day 2
  Continuous variable to be assessed as : Narcotics requested by the patient and administered post-procedural day 1 and day 2 (Total and separately assessed). All narcotics will be converted to IV morphine equianalgesic equivalent conversion factors according to American Pain Society
Incident of oral Morbidities related to the procedure | intraoperative up to 1 month post-procedure
  Event rate nominal variable to be assessed as: oral morbidity post-procedure categorized according to Clavien Dindo-Classification

SECONDARY OUTCOMES:
Post-operative Pain score | Post-op day 2
  Continuous variables to be assessed as: Post-operative oral pain score measured using 10 point visual analogue score for pain assessment (minimum 0 or no pain to maximum 10 most painful)
Post-operative Pain score | Post-op day 3
  Continuous variables to be assessed as: Post-operative oral pain score measured using 10 point visual analogue score for pain assessment (minimum 0 or no pain to maximum 10 most painful)
Post-operative Pain score | Post-op day 1 month follow-up
  Continuous variables to be assessed as: Post-operative oral pain score measured using 10 point visual analogue score for pain assessment (minimum 0 or no pain to maximum 10 most painful)
number of participants with return to regular diet post-procedure | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)
Incident of post-procedural peri-oral numbness | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)
Incident of post-procedural salivary changes | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (more, less or none)
Incident of post-procedural taste changes | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)
Incident of post-procedural speech changes | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)
Number of participants with post-procedure full-mouth opening | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)
Number of participants report perceived adverse effect related to local anesthetics | Post-op day 1- 3, then 1 month follow-up (Optional daily up to post-op day 7 and monthly after 1 month up to one year or beyond)
  Event rate nominal variable to be assessed using survey question (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt McCammon, MD FACS, Principal Investigator — Eastern Virginia Medical School- Urology
Locations (1):
- Urology of Virginia, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chua ME, Zuckerman JM, Strehlow R 6th, Virasoro R, DeLong JM, Tonkin J, McCammon KA. Liposomal Bupivacaine Local Infiltration for Buccal Mucosal Graft Harvest Site Pain Control: A Single-blinded Randomized Controlled Trial. Urology. 2020 Nov;145:269-274. doi: 10.1016/j.urology.2020.06.067. Epub 2020 Jul 18. PMID 32692990